CLINICAL TRIAL: NCT06445179
Title: Robot-Assisted Versus Standard Laparoscopic Approach of Total Hysterectomy for Deep Infiltrating Endometriosis and Adenomyosis: A Multicenter, Open-label Randomized Controlled Trial
Brief Title: ENDOmetriosis Robotic Assisted Surgery
Acronym: ENDO-RAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A00350-47
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized into two parallel groups.
Masking Description: The ENDO-RAS Trial is a multicenter, randomized, controlled, and open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without Robotic-Assisted (Active Comparator): In the control group, all patients will undergo a Total Laparoscopic Hysterectomy. The number of ports needed for the laparoscope and assistants will be reported.
  Interventions: Procedure: Total Laparoscopic Hysterectomy; Device: Ureterolysis
- Robotic-Assisted (Experimental): All patients in the experimental group will undergo a Robotic-Assisted Total Laparoscopic Hysterectomy using either the HugoTM Robot-Assisted Surgery system (Medtronic©), the Da Vinci® Xi or X Surgical System, or CMR versus (if available). The number of ports required for the laparoscope, robotic arms, and assistants will be documented.
  Interventions: Procedure: Total Laparoscopic Hysterectomy; Device: Ureterolysis

INTERVENTIONS:
Procedure: Total Laparoscopic Hysterectomy — The standard procedure for performing total hysterectomy will also follow the Querleu and Morrow classification system, which divides the procedure into four types based on the extent of resection:
  * Type A: minimum resection of paracervix.
  * Type B: transection of the paracervix and the ureter.
  * Type C: Transection of paracervix at the junction with the internal iliac vascular system
  * Type D: Laterally extended resection. Furthermore, bilateral ureterolysis will be performed with the option of bilateral concomitant salpingo-oophorectomy.
Device: Ureterolysis — unilateral or bilateral ureterolysis with or without bilateral adnexectomy

SUMMARY:
The purpose of this study is to compare the robot-assisted approach with the laparoscopic approach in terms of reducing the rates of intraoperative and postoperative complications in patients undergoing total hysterectomy for DIE and adenomyosis without digestive tract involvement.

DETAILED DESCRIPTION:
The ENDO-RAS trial aims to evaluate the safety and effectiveness of robot-assisted laparoscopy compared to conventional laparoscopy for hysterectomy in patients with Deep infiltrating endometriosis and adenomyosis without digestive tract involvement, as verified by magnetic resonance imaging and classified using both the ENZIAN and Deep Pelvic Endometriosis Index classifications. These classifications are used to evaluate Deep infiltrating endometriosis and reproducibly predict the occurrence of postoperative complications.

Eligible patients will be recruited from the gynecological surgery department after meeting the inclusion and non-inclusion criteria and signed informed consent forms. Participants will then be randomly assigned to receive either robot-assisted total laparoscopic hysterectomy or total laparoscopic hysterectomy.

The ENDO-RAS Trial is a multicenter, randomized, controlled, and open-label study. Eligible patients will be randomized into two parallel groups.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Diagnosed adenomyosis, either internal or external (magnetic resonance imaging) per the Enzian and dPEI classifications.
* Diagnosed deep infiltrating endometriosis per the Enzian and dPEI classifications, without the involvement of the digestive tract.
* Failure of first- and second-line medical treatment.
* Eligibility for total hysterectomy with complete removal of endometriosis lesions.
* Participants covered by entitled to social security.
* All participants must provide written informed consent before undergoing the surgical procedure.

Exclusion Criteria:

* Digestive tract involvement.
* Adenomyosis only.
* Contraindications to surgery.
* Participants who are under guardianship, curatorship, or deprivation of liberty.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Intra and post-operative complication rates | 3 months
  Rate of intra- and post-operative complications (Clavien-Dindo grade 2 or higher) following surgery (Total Laparoscopic Hysterectomy).

SECONDARY OUTCOMES:
Short Form Health Survey (SF-36) | At baseline and at 3, 6, and 12 month.
  Patients' quality of life COmpletion of hte Endometriosis-related quality of life
Patients' sexual quality of life | At baseline and at 3, 6, and 12 months.
  Completion of the Sexual quality-of-life using the Female Sexual Function Index (FSFI) A 19-point questionnaire with a scale from 0 to 5.
Duration of the intervention | Time from incision to closure (12 months)
  The mean operative time (minutes) which will be defined as the time from incision to closure.
Intraoperative and postoperative complications | At 1, 6, and 12 months
  Rate of intraoperative and postoperative complications, according to the Clavien-Dindo classification
Blood loss | During the intervention
  Volume of blood loss (mL)
Pain symptoms | At 30 days, and at 3, 6, and 12 months postoperatively.
  Mean numeric rating scale (NRS) from 0 to 10 where 10 is extreme pain.
Length of hospital stay | From the intervanetion day to the day of discharge from hospital (within 30 days after surgery)
  Total number of days in the hospital
Hospital readmissions | 30 days after surgery
  Rate of hospital readmissions
Reoperation | Within 30 days after surgery
  Rate of reoperation
Robotic and complex laparoscopic expertise of the surgeons | 1 year
  Number of robotic and complex laparoscopic procedures performed by the surgeons involved and in the hospitals involved
Completion of Questionnaires Borg CR-10 Scale | Day 0 (surgery)
  Perceived exertion by surgeons of laparoscopic and robotic intervention.
Endometriosis Health Profile-30 (EHP30) | At baseline and at 3, 6, and 12 month.
  Patients' quality of life COmpletion of hte Endometriosis-related quality of life
Completion of Questionnaires NASA-TLX | Day 0 (surgery)
  Perceived exertion by surgeons of laparoscopic and robotic intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Privé de Provence, Aix-en-Provence
  - Hôpital Privé le Bois, Lille

IPD SHARING:
Plan to Share IPD: Yes
Only data that is strictly relevant and directly used in the published article will be eligible for sharing. No data outside the scope of the published analysis will be transmitted.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting from 2028 for one year
Access Criteria: Data will be made available upon reasonable request from the journal of the published article, strictly for reanalysis of the published results. In such instances, requests should be directed via email to the corresponding author. The statistical code employed for the original analyses may also be shared if deemed necessary. Depending on the nature of the request, the original authors may be invited to participate in the reanalysis.
  Data will be shared in the form of an anonymized Excel file, in full compliance with applicable data protection regulations. No information will permit the direct or indirect identification of patients. The shared data may only be used for the specific purpose defined in the initial request. No secondary use or data transfer agreement will be considered or negotiated. Please let us know if any further clarification is required.

REFERENCES:
- [Derived] Renso M, Bendifallah S, Estrade JP, Merlot B, Roman H, Vidal F, Collinet P. Robot-assisted versus standard laparoscopic approach of total hysterectomy for deep infiltrating endometriosis and adenomyosis (ENDORAS TRIAL): study protocol for a randomised controlled trial. BMJ Open. 2025 Nov 28;15(11):e108125. doi: 10.1136/bmjopen-2025-108125. PMID 41314847